CLINICAL TRIAL: NCT06706869
Title: A PHASE 1, OPEN-LABEL, 2-PART STUDY TO ESTIMATE SEPARATELY THE EFFECT OF ITRACONAZOLE AND FOOD ON THE PHARMACOKINETICS OF PF-07258669 IN OLDER ADULT OR HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn if the Study Medicine Called Itraconazole and if Food Changes How the Body Processes the Other Study Medicine Called PF 07258669 in Older Adults or Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C4541012
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Masking Description: Parts A and B are not masked. Part A is not randomized. Part B is randomized to Sequence 1 or Sequence 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Period 1 (Experimental): A single oral dose of PF-07258669 on Study Day 1
  Interventions: Drug: PF-07258669
- Part A: Period 2 (Experimental): Itraconazole QD orally on Study Days 4 to 11. PF-07258669 will be co administered on Study Day 7.
  Interventions: Drug: PF-07258669; Drug: Itraconazole
- Part B: Sequence 1 (Experimental): A single oral dose of PF-07258669 on Study Days 1 and 4 under fasted and fed conditions respectively.
  Interventions: Drug: PF-07258669
- Part B: Sequence 2 (Experimental): A single oral dose of PF-07258669 on Study Days 1 and 4 under fed and fasted conditions respectively.
  Interventions: Drug: PF-07258669

INTERVENTIONS:
Drug: PF-07258669 — Tablet
Drug: Itraconazole — Solution
  Arms: Part A: Period 2

SUMMARY:
The purpose of this study is to learn how the medicine called itraconazole and food changes how the body processes another study medicine called PF-07258669 in older adults or healthy adults.

The study medicine PF-07258669 is developed for the treatment of unintended weight loss in older adults. People with this condition have decreased appetite and food intake, which is an important reason for poor nutrition and health results in people with unintended weight loss. The study has two parts: Part A and Part B.

The study is seeking participants who:

1. Are males or females who can no longer have children.
2. Part A Only: Are at least 65 years old and in reasonably good health. Part B Only: Are at least 18 years old and in good health.
3. Part A Only: Have a body mass index (BMI) of 16 to 27 kilogram per meter squared and a total body weight of more than 40 kilograms (88 pounds). Part B Only: Have a BMI of 16-32 kilogram per meter squared and a total body weight of more than 50 kilograms (110 pounds).

For Part A: Participants will take the study medicine PF-07258669 as tablets by mouth once on Day 1 at the study clinic and stay at the clinic for about 12 days. Then starting on Day 4, participants will take itraconazole as liquid by mouth for eight days. On Day 7, itraconazole will be taken together with PF-07258669.

For Part B: Participants will take the study medicine PF-07258669 as tablets by mouth once on Day 1 without breakfast at the study clinic and stay at the clinic for about 7 days. On Day 4, participant will take the study medicine after breakfast. A different group of participants will follow a similar procedure, but they will take the medicine after breakfast on Day 1 and without breakfast on Day 4.

For Parts A and B: At the clinic, the study team will observe the participants and take urine and blood samples to look at the levels of PF-07258669. The participants will receive a follow up telephone call about one month later.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who can no longer have children.
2. Part A Only: At least 65 years old. Part B Only: At least 18 years old.
3. In reasonably good health.
4. Part A Only: Body mass index (BMI) of 16-27 kg/m2; and a total body weight >40 kg (88 lb.). Part B Only: BMI of 16-32 kg/m2; and a total body weight >50 kg (110 lb.).

Exclusion criteria

1. Evidence or history of clinically significant medical conditions.
2. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb).
3. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
4. Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Baseline to Day 12 (Part A); Baseline to Day 7 (Part B)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Baseline to Day 12 (Part A); Baseline to Day 7 (Part B)
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) [if data permit, otherwise AUClast] | Baseline to Day 12 (Part A); Baseline to Day 7 (Part B)

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events | Baseline to Day 46 (Part A); Baseline to Day 39 (Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Research Centers of America, Hollywood, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4541012